CLINICAL TRIAL: NCT01992523
Title: Mojito Study (Mashed Or Just Integral Pill of TicagrelOr ? )
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: David Antoniucci (Other)
Collaborators: AstraZeneca (Industry); A.R. CARD Onlus Foundation (Other)
Responsible Party: Sponsor-Investigator, David Antoniucci, Director, Division of Invasive Cardiology, Careggi Hospital
Organization: Careggi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOJITO Study
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Acute Coronary Syndrome; Adverse Reaction to Antiplatelet Agent
Keywords: Ticagrelor; antiplatelet; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor mashed pills (Experimental): Ticagrelor loading dose (LD) 180 mg as mashed pills
  Interventions: Drug: Ticagrelor mashed pills
- Ticagrelor integral pills (Active Comparator): Ticagrelor loading dose (LD) 180 mg as integral pills
  Interventions: Drug: Ticagrelor integral pills

INTERVENTIONS:
Drug: Ticagrelor mashed pills — The loading dose will be performed as soon as possible in the Emergency Room or in the Cath Lab. In all case before the end of the PCI (percutaneous coronary intervention) . In the case of vomit in the first hour after drug loading dose a new reduced loading dose will be administered (90 mg Ticagrelor). Mashed pills administration will be prepared placing 2 ticagrelor pills in a mortar and mashing for 60 seconds using a pestle. The total contents of the mortar will be transferred to the dosing cup, 50 mL of purify water will be added, and the suspension mixed up before drinking. Afterwards, 100 mL of purify water will be administered to the patient.
  Arms: Ticagrelor mashed pills
Drug: Ticagrelor integral pills — The loading dose will be performed as soon as possible in the Emergency Room or in the Cath Lab. In all case before the end of the PCI (percutaneous coronary intervention) . In the case of vomit in the first hour after drug loading dose a new reduced loading dose will be administered (90 mg Ticagrelor).
  Arms: Ticagrelor integral pills

SUMMARY:
The aim of the Mashed Or Just Integral pill of TicagrelOr (MOJITO) study is to evaluate the superiority of Ticagrelor 180 mg LD mashed pill versus Ticagrelor 180 mg LD integral pill both orally administrated in decreasing residual platelet reactivity 1 hour after the administration among 70 patients with STEMI (ST segment elevation myocardial infarction) undergoing PPCI (primary percutaneous coronary intervention) with bivalirudin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting within 12 hours from the onset of symptoms with STEMI
* Informed, written consent

Exclusion Criteria:

* Age < 18 years or Age > 75 years
* Active bleeding; bleeding diathesis; coagulopathy
* Increased risk of bradycardiac events
* History of gastrointestinal or genitourinary bleeding <2 months
* Major surgery in the last 6 weeks
* History of intracranial bleeding or structural abnormalities
* Suspected aortic dissection
* Any other condition that may put the patient at risk or influence study results or investigator's opinion (severe hemodynamic instability, known malignancies or other comorbid conditions with life expectancy <1 year)
* Administration in the week before the index event of clopidogrel, ticlopidine, prasugrel, ticagrelor, thrombolytics, bivalirudin, low-molecular weight heparin or fondaparinux .
* Concomitant oral or IV therapy with strong CYP3A inhibitors or strong CYP3A inducers, CYP3A with narrow therapeutic windows
* Known relevant hematological deviations: Hb <10 g/dl, Thrombi. <100x10^9/l
* Use of coumadin derivatives within the last 7 days
* Chronic therapy with ticagrelor, prasugrel, clopidogrel or ticlopidine
* Known severe liver disease, severe renal failure
* Known allergy to the study medications
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Parodi, MD, Principal Investigator — Careggi Hospital, Division of Invasive Cardiology; David Antoniucci, MD, Study Director — Careggi Hospital, Division of Invasive Cardiology
Locations (2):
- Department of Cardiology, Patras University Hospital, Pátrai, Greece
- Careggi Hospital, Florence, Italy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ticagrelor Mashed Pills | Ticagrelor Integral Pills
Started | 41 | 41
Completed | 41 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor Mashed Pills | Ticagrelor Integral Pills | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (13) | 61 (14) | 62 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 31 | 33 | 64
Region of Enrollment [Number; unit: participants]
  Greece | 15 | 15 | 30
  Italy | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Residual Platelet Reactivity
Description: residual platelet reactivity by Platelet Reactivity Units (PRU) VerifyNow 1 hour after ticagrelor LD.
Time Frame: 1 hour
Population: Continuous data were expressed as mean ± standard deviation or medians (quartiles) as appropriate, and categorical data as proportions (%). A P value < .05 was considered statistically significant. All tests were two-sided.
Measure: Median (Inter-Quartile Range); unit: PRU (P2Y12 reaction units)
Arm/Group | Ticagrelor Mashed Pills | Ticagrelor Integral Pills
Number analyzed (Participants) | 41 | 41
PRU (P2Y12 reaction units) | 168 [61 to 251] | 252 [167 to 301]
Statistical Analysis 1: Comparison: Ticagrelor Mashed Pills vs Ticagrelor Integral Pills; Continuous data were expressed as mean ± standard deviation or medians (quartiles) as appropriate, and categorical data as proportions (%). Data were compared by means of the chi-2 test or Fisher exact test for categorical variables and unpaired t test or Mann-Whitney U-test for continuous variables, as appropriate. A P value < .05 was considered statistically significant. All tests were two-sided; Test type: Superiority or Other; p = 0.006, t-test, 2 sided

2. Secondary Outcome: High Residual Platelet Reactivity
Description: The percent of patients with a high residual platelet reactivity (PRU > 208) 1 hour after ticagrelor LD.
Time Frame: 1 hour
Population: Categorical data were expressed as proportions (%)
Measure: Number; unit: percentage of partecipants
Arm/Group | Ticagrelor Mashed Pills | Ticagrelor Integral Pills
Number analyzed (Participants) | 41 | 41
percentage of partecipants | 35 | 63

3. Secondary Outcome: Bleeding Events
Description: Percentage of participants with Major, minor, minimal bleeding (TIMI criteria) events
Time Frame: 48 hours
Measure: Number; unit: percentage of partecipants
Arm/Group | Ticagrelor Mashed Pills | Ticagrelor Integral Pills
Number analyzed (Participants) | 41 | 41
percentage of partecipants | 2.4 | 7

4. Secondary Outcome: Dyspnoea and/or Symptomatic Bradycardia
Description: Percentage of participants with Occurrence of dyspnoea and/or symptomatic bradycardia
Time Frame: 6 months
Population: Continuous data were expressed as mean ± standard deviation or medians (quartiles) as appropriate, and categorical data as proportions (%)
Measure: Number; unit: percentage of partecipants
Arm/Group | Ticagrelor Mashed Pills | Ticagrelor Integral Pills
Number analyzed (Participants) | 41 | 41
percentage of partecipants | 12 | 12

ADVERSE EVENTS:
Time Frame: Intra-hospital events
Groups:
- Ticagrelor Mashed Group: patients taking orally 180 mg ticagrelor mashed tablets
- Ticagrelor Integral Group: patients taking orally 180 mg ticagrelor integral tablets
Arm/Group | Ticagrelor Mashed Group | Ticagrelor Integral Group
Serious Adverse Events (participants affected / at risk) | 2/41 | 2/41
Other Adverse Events (participants affected / at risk) | 9/41 | 8/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor Mashed Group (N=41) | Ticagrelor Integral Group (N=41)
death (Cardiac disorders) | 1 (1) | 1 (1) — Cardiovascular and non cardiovascular death
Re-infarction (Cardiac disorders) | 1 (1) | 0 (0)
stroke (Vascular disorders) | 0 (0) | 0 (0)
Major bleeding (TIMI criteria) (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor Mashed Group (N=41) | Ticagrelor Integral Group (N=41)
TIMI minor bleeding (TIMI criteria) (Vascular disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Ventricular pauses >= 3 sec (Cardiac disorders) | 0 (0) | 1 (1)
Serum creatinine increase (Renal and urinary disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No